CLINICAL TRIAL: NCT05870865
Title: A Randomized, Double-Blind, Vehicle-Controlled, Phase 2 Trial to Evaluate the Anti-pruritic Efficacy, Safety, Tolerability, and Pharmacokinetics of ASN008 in Adults With Mild to Moderate Atopic Dermatitis
Brief Title: A Study to Evaluate the Anti-pruritic Effectiveness of ASN008 in Adults With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Formation Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASN008-201
Record Dates: First submitted 2023-03-30; First posted 2023-05-23 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Dermatitis, Atopic; Pruritus
Keywords: Dermatitis, Atopic; Pruritus; Eczema; Itch
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus; Eczema

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized to 1 of 4 cohorts: ASN008 gel 1.25 percent, 2.5 percent, 5 percent, or matching vehicle.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: At all times, treatment and randomization information will be kept confidential and will not be released to the Sponsor's trial team until database lock is completed. Investigators, participants, and clinical staff will remain blinded throughout the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ASN008 1.25% (Experimental): ASN008 1.25% twice daily topical application applied as a thin layer (approximately 2 mg/cm^2) for 4 weeks (28 days)
  Interventions: Drug: ASN008
- ASN008 2.5% (Experimental): ASN008 2.5% twice daily topical application applied as a thin layer (approximately 2 mg/cm^2) for 4 weeks (28 days)
  Interventions: Drug: ASN008
- ASN008 5% (Experimental): ASN008 5% twice daily topical application applied as a thin layer (approximately 2 mg/cm^2) for 4 weeks (28 days)
  Interventions: Drug: ASN008
- ASN008 Matching Vehicle (Placebo Comparator): ASN008 matching vehicle twice daily topical application applied as a thin layer (approximately 2 mg/cm^2) for 4 weeks (28 days)
  Interventions: Other: ASN008 Matching Vehicle

INTERVENTIONS:
Drug: ASN008 — ASN008 topical gel applied twice daily.
  Arms: ASN008 1.25%; ASN008 2.5%; ASN008 5%
Other: ASN008 Matching Vehicle — The ASN008 matching vehicle formulation matches the formulation of each ASN008 topical gel dose, but contains no ASN008.
  Arms: ASN008 Matching Vehicle

SUMMARY:
The goal of this clinical trial is to evaluate ASN008 in people with itch caused by eczema. The main questions it aims to answer are:

* What is the efficacy and safety of ASN008?
* What is the impact of ASN008 on itch in patients with atopic dermatitis? Participants will be asked to apply topical ASN008, or matching vehicle (placebo containing no active drug), to their eczema lesions twice daily for 4 weeks.

Researchers will compare 3 different doses of ASN008 and a matching vehicle group to see which group responds best.

DETAILED DESCRIPTION:
All participants will sign an informed consent form and undergo screening (within 28 days prior to Day 1). During the screening period, all treatments for Atopic Dermatitis (AD) (also known as eczema) and/or itch will be stopped to allow for wash out, as applicable and according to eligibility requirements. Consistent daily or twice daily use of a non-prescription emollient is required at least 7 days prior to Day 1 and throughout the trial until the follow-up (Week 8). No other products, including, but not limited to, topical corticosteroids, calcineurin inhibitors, biologics, or Janus Kinase (JAK) inhibitors (topical or oral) may be used during the trial.

Eligible participants will be randomized in a 1:1:1:1 ratio to receive ASN008 gel 1.25 percent, ASN008 gel 2.5 percent, ASN008 gel 5.0 percent, or matching vehicle twice daily for 4 weeks (28 days), followed by a 4-week (28-day) follow-up period. The first dose of study treatment will be applied on Day 1 and the last dose will be applied on the morning of Day 28.

Participants will be required to participate in 8 scheduled visits: Screening; Randomization (remote visit); Day 1; Week 1 (Day 8); Week 2 (Day 15); Week 3 (Day 22); Week 4 (Day 28); and Week 8 (Day 56)/early termination (ET).

The trial duration per participant is up to 12 weeks (84 days): including up to 4 weeks (28 days) for the screening period, 4 weeks (28 days) for the treatment period, and up to 4 weeks (28 days) for the follow-up period.

A participant is considered to have reached the end of the trial when they have completed their Day 56 (Week 8) or ET visit. The trial will be considered complete when the last participant has completed their last trial visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, 18 years or older, at the time of informed consent.
* Diagnosis of mild to moderate AD for at least 12 months with no significant disease flares for at least 4 weeks before Screening (based upon medical chart, treating physician, or participant report with documented clinical confirmation by the Investigator)
* Validated Investigator Global Assessment (vIGA) score of 2 or 3 at Day 1.
* Body surface area (BSA) affected by AD ≤20% at Day 1.
* Peak Pruritus NRS ≥7 at Day 1.
* Body mass index (BMI) ≤40 kg/m2 at Screening.
* Willingness to avoid pregnancy or fathering children.
* Participant is willing to participate for the duration of the trial, comply with all trial procedures, and is capable of giving informed consent.

Exclusion Criteria:

* Any female who is breastfeeding, pregnant, or who is planning to become pregnant during the trial.
* Active infection requiring treatment, including skin infections (including clinically infected AD).
* History of skin disease or presence of a skin condition that, in the opinion of the Investigator, would interfere with trial assessments.
* Any clinically significant medical or psychiatric condition or physical/laboratory/ECG/vital signs abnormality that would, in the opinion of the Investigator, put the participant at undue risk or interfere with interpretation of trial results.
* Use of any of the following treatments within the indicated washout period before Day 1:

  1. Doxepin, hydroxyzine, or diphenhydramine use within 1 week prior to Day 1.
  2. Use of topical product containing urea or any antihistamine within 1 week prior to Day 1.
  3. Use of systemic antibiotic within 2 weeks, or topical antibiotics within 1 week, prior to Day 1.
  4. Atopic dermatitis topical medication use within 2 weeks prior to Day 1, including, but not limited to, topical corticosteroids, crisaborole and any other topical phosphodiesterase-4 inhibitor, calcineurin inhibitors, JAK inhibitors, tars, bleach, antimicrobials, medical devices, and bleach or oatmeal baths.
  5. Psoralen-UV-A or UV-B phototherapy (including tanning beds) or excimer laser within 4 weeks prior to Day
  6. Systemic medication use including biologics that could affect AD less than 6 weeks prior to Day 1 (e.g., retinoids, calcineurin inhibitors, methotrexate, cyclosporine, hydroxycarbamide [hydroxyurea], azathioprine, oral/injectable corticosteroids), biologics and JAK inhibitors.
* Known hypersensitivity to ASN008 or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - TrialSpark Investigative Site 0106, Scottsdale, Arizona
  - TrialSpark Investigative Site 0118, Hot Springs, Arkansas
  - TrialSpark Investigative Site 0123, Beverly Hills, California
  - TrialSpark Investigative Site 0113, Fremont, California
  - TrialSpark Investigative Site 0101, Los Angeles, California
  - TrialSpark Investigative Site 0103, Miami Lakes, Florida
  - TrialSpark Investigative Site 0129, Miramar, Florida
  - TrialSpark Investigative Site 0131, Clarksville, Indiana
  - TrialSpark Investigative Site 0109, Indianapolis, Indiana
  - TrialSpark Investigative Site 0112, Louisville, Kentucky
  - TrialSpark Investigative Site 0108, Baton Rouge, Louisiana
  - TrialSpark Investigative Site 0124, Monroe, Louisiana
  - TrialSpark Investigative Site 0107, Auburn Hills, Michigan
  - TrialSpark Investigative Site 0102, Saint Joseph, Missouri
  - TrialSpark Investigative Site 0115, Kew Gardens, New York
  - TrialSpark Investigative Site 0119, New York, New York
  - TrialSpark Investigative Site 0105, Wilmington, North Carolina
  - TrialSpark Investigative Site 0125, Mason, Ohio
  - TrialSpark Investigative Site 0127, Oklahoma City, Oklahoma
  - TrialSpark Investigative Site 0122, Philadelphia, Pennsylvania
  - TrialSpark Investigative Site 0121, Houston, Texas
  - TrialSpark Investigative Site 0130, Pflugerville, Texas
  - TrialSpark Investigative Site 0114, San Antonio, Texas
  - TrialSpark Investigative Site 0126, San Antonio, Texas
  - TrialSpark Investigative Site 0110, Springville, Utah
  - TrialSpark Investigative Site 0117, Richmond, Virginia
  - TrialSpark Investigative Site 0128, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Randomized
Arm/Group | ASN008 1.25% | ASN008 2.5% | ASN008 5% | ASN008 Matching Vehicle
Started | 36 | 36 | 36 | 36
Completed | 34 | 32 | 32 | 33
Not Completed | 2 | 4 | 4 | 3
Not completed — Did not receive study treatment | 2 | 4 | 4 | 3
Period: Treatment Period
Arm/Group | ASN008 1.25% | ASN008 2.5% | ASN008 5% | ASN008 Matching Vehicle
Started | 34 | 32 | 32 | 33
Completed | 33 | 29 | 28 | 30
Not Completed | 1 | 3 | 4 | 3
Not completed — Adverse Event | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | ASN008 1.25% | ASN008 2.5% | ASN008 5% | ASN008 Matching Vehicle | Total
Number analyzed (Participants) | 34 | 32 | 32 | 33 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 31 | 29 | 28 | 117
  >=65 years | 5 | 1 | 3 | 5 | 14
Age, Continuous [Least Squares Mean (Standard Deviation); unit: years] | 47.7 (15.45) | 41.8 (12.54) | 43.3 (15.95) | 46.5 (16.04) | 44.9 (15.09)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 14 | 15 | 7 | 10 | 46
  Female | 20 | 17 | 25 | 23 | 85
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity : Hispanic or Latino | 14 | 11 | 15 | 11 | 51
  Ethnicity : Not Hispanic or Latino | 20 | 21 | 17 | 22 | 80
  Race: White | 25 | 19 | 23 | 22 | 89
  Race: Black or African American | 8 | 11 | 7 | 11 | 37
  Race: Asian | 0 | 2 | 1 | 0 | 3
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Race: Other | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Daily Peak Pruritus Numerical Rating Scale (NRS)
Description: Percent change of 7-day average daily peak pruritus NRS from Baseline to Week 4
Time Frame: Baseline to Week 4
Population: Modified Intent to Treat
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | ASN008 1.25% | ASN008 2.5% | ASN008 5% | ASN008 Matching Vehicle
Number analyzed (Participants) | 30 | 30 | 26 | 31
percent change | -45.6 (5.04) | -55.8 (5.13) | -48.3 (5.2) | -49.9 (4.99)
Statistical Analysis 1: Comparison: ASN008 1.25% vs ASN008 Matching Vehicle; Test type: Superiority; p = 0.5483, Mixed Models Analysis; Mean Difference (Final Values) = 4.28
Statistical Analysis 2: Comparison: ASN008 2.5% vs ASN008 Matching Vehicle; Test type: Superiority; p = 0.4123, Mixed Models Analysis; Mean Difference (Final Values) = -5.89
Statistical Analysis 3: Comparison: ASN008 5% vs ASN008 Matching Vehicle; Test type: Superiority; p = 0.8177, Mixed Models Analysis; Mean Difference (Final Values) = 1.66

2. Secondary Outcome: Pruritus Response of ASN008 Topical Gel on Atopic Dermatitis (AD) Assessed by Daily Peak Pruritus NRS
Description: Pruritus response defined as 7-day average of daily peak pruritus NRS reduction greater than or equal to 4 points from Baseline to Week 4
Time Frame: Baseline to Week 4
Population: Modified Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | ASN008 1.25% | ASN008 2.5% | ASN008 5% | ASN008 Matching Vehicle
Number analyzed (Participants) | 34 | 32 | 32 | 33
Participants | 12 | 22 | 15 | 15
Statistical Analysis 1: Comparison: ASN008 1.25% vs ASN008 Matching Vehicle; Test type: Superiority; p = 0.4601, Fisher Exact; Odds Ratio (OR) = 0.66
Statistical Analysis 2: Comparison: ASN008 2.5% vs ASN008 Matching Vehicle; Test type: Superiority; p = 0.0804, Fisher Exact; Odds Ratio (OR) = 2.64
Statistical Analysis 3: Comparison: ASN008 5% vs ASN008 Matching Vehicle; Test type: Superiority; p > 0.9999, Fisher Exact; Odds Ratio (OR) = 1.06

3. Secondary Outcome: Mean Change From Baseline in Eczema Area and Severity Index (EASI) Score
Description: This outcome measure evaluates the change and percent change in the Eczema Area and Severity Index (EASI) score from Baseline to Week 4. The EASI score measures the extent and severity of eczema across four body regions: head/neck, trunk, upper limbs, and lower limbs. Two components are assessed: severity of erythema, edema/papulation, excoriation, and lichenification (each scored 0 to 3, with 0 = none and 3 = severe) and the surface area affected (scored 0 to 6, with 0 = no involvement and 6 = 90%-100% involvement).
  Subscale scores are combined using weighted multipliers for each region (head/neck 0.1, upper limbs 0.2, trunk 0.3, lower limbs 0.4) to calculate the total score. The EASI is a composite score ranging from 0 (no eczema) to 72 (maximum severity and extent). Scores are summed to account for the severity of lesions and the percentage of body surface area (BSA) affected in each region.
Time Frame: Baseline to Week 4
Population: Modified Intent to Treat
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ASN008 1.25% | ASN008 2.5% | ASN008 5% | ASN008 Matching Vehicle
Number analyzed (Participants) | 32 | 28 | 25 | 30
score on a scale | -2.7 (0.40) | -3.5 (0.43) | -2.6 (0.45) | -3.4 (0.41)
Statistical Analysis 1: Comparison: ASN008 1.25% vs ASN008 Matching Vehicle; Test type: Superiority; p = 0.2146, Mixed Models Analysis; Mean Difference (Final Values) = 0.72
Statistical Analysis 2: Comparison: ASN008 2.5% vs ASN008 Matching Vehicle; Test type: Superiority; p = 0.8851, Mixed Models Analysis; Mean Difference (Final Values) = -0.09
Statistical Analysis 3: Comparison: ASN008 5% vs ASN008 Matching Vehicle; Test type: Superiority; p = 0.1835, Mixed Models Analysis; Mean Difference (Final Values) = 0.81

4. Secondary Outcome: Mean Change From Baseline in Total Body Surface Area (BSA)
Description: Change from Baseline in total BSA at week 4.
Time Frame: Baseline to Week 4
Population: Modified Intent to Treat
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | ASN008 1.25% | ASN008 2.5% | ASN008 5% | ASN008 Matching Vehicle
Number analyzed (Participants) | 32 | 28 | 25 | 30
Percentage | -2.6 (0.56) | -2.9 (0.59) | -1.5 (0.60) | -2.4 (0.56)
Statistical Analysis 1: Comparison: ASN008 1.25% vs ASN008 Matching Vehicle; Test type: Superiority; p = 0.7982, Mixed Models Analysis; Mean Difference (Final Values) = -0.2
Statistical Analysis 2: Comparison: ASN008 2.5% vs ASN008 Matching Vehicle; Test type: Superiority; p = 0.5640, Mixed Models Analysis; Mean Difference (Final Values) = -0.5
Statistical Analysis 3: Comparison: ASN008 5% vs ASN008 Matching Vehicle; Test type: Superiority; p = 0.2939, Mixed Models Analysis; Mean Difference (Final Values) = 0.9

5. Secondary Outcome: Mean Change From Baseline in the Patient-Oriented Eczema Measure (POEM)
Description: This outcome measure evaluates the change in the the Patient-Oriented Eczema Measure (POEM) score from Baseline to Week 4.The POEM is a self-assessment tool that evaluates eczema severity based on patient-reported symptoms over the previous week. It includes 7 questions addressing common symptoms: itch, sleep disturbance, bleeding, weeping, cracking, flaking, and dryness. Each question is scored on a scale from 0 to 4 based on frequency (0 = no days, 1 = 1-2 days, 2 = 3-4 days, 3 = 5-6 days, 4 = every day). The scores are summed to generate a total score ranging from 0 to 28. Scores are interpreted as follows: 0-2 = clear or almost clear, 3-7 = mild eczema, 8-16 = moderate eczema, 17-24 = severe eczema, and 25-28 = very severe eczema. Higher scores indicate a greater symptom burden and worse disease severity.
Time Frame: Baseline to Week 4
Population: Modified Intent to Treat
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ASN008 1.25% | ASN008 2.5% | ASN008 5% | ASN008 Matching Vehicle
Number analyzed (Participants) | 31 | 28 | 25 | 29
score on a scale | -5.0 (1.04) | -7.8 (1.08) | -6.3 (1.11) | -6.4 (1.06)
Statistical Analysis 1: Comparison: ASN008 1.25% vs ASN008 Matching Vehicle; Test type: Superiority; p = 0.3579, Mixed Models Analysis; Mean Difference (Final Values) = 1.4
Statistical Analysis 2: Comparison: ASN008 2.5% vs ASN008 Matching Vehicle; Test type: Superiority; p = 0.3466, Mixed Models Analysis; Mean Difference (Final Values) = -1.4
Statistical Analysis 3: Comparison: ASN008 5% vs ASN008 Matching Vehicle; Test type: Superiority; p = 0.9527, Mixed Models Analysis; Mean Difference (Final Values) = 0.1

6. Other Pre Specified Outcome: Inter- and Intra-subject Variability of ASN008 Pharmacokinetics (PK) Characterized by Peak Plasma Concentration (Cmax)
Description: ASN008 PK will be characterized using population-based methods to include Peak Plasma Concentration (Cmax).
Time Frame: Baseline and Week 4
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Inter- and Intra-subject Variability of ASN008 Pharmacokinetics Characterized by Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: ASN008 PK will be characterized using population-based methods to include area under the plasma concentration versus time curve (AUC)
Time Frame: Baseline and Week 4
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: Number of participants who experienced a TEAE.
Time Frame: Baseline to Day 56
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | ASN008 1.25% | ASN008 2.5% | ASN008 5% | ASN008 Matching Vehicle
Number analyzed (Participants) | 34 | 32 | 32 | 33
Participants | 12 | 14 | 11 | 8

9. Other Pre Specified Outcome: Number of Investigational Product (IP)-Related TEAEs
Description: Number of participants who experienced an IP-related TEAE.
Time Frame: Baseline to Day 56
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | ASN008 1.25% | ASN008 2.5% | ASN008 5% | ASN008 Matching Vehicle
Number analyzed (Participants) | 34 | 32 | 32 | 33
Participants | 1 | 3 | 3 | 1

10. Other Pre Specified Outcome: Incidence of TEAEs Leading to Treatment Discontinuation
Description: Incidence of TEAEs leading to treatment discontinuation from first dose through completion of follow-up period (up to a maximum of 56 days)
Time Frame: Baseline to Day 56
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | ASN008 1.25% | ASN008 2.5% | ASN008 5% | ASN008 Matching Vehicle
Number analyzed (Participants) | 34 | 32 | 32 | 33
Participants | 1 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected beginning after participant enrollment, before treatment, during treatment, and up to 28 days following the cessation of treatment, up to Day 56/Week 8.
Arm/Group | ASN008 1.25% | ASN008 2.5% | ASN008 5% | ASN008 Matching Vehicle
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/32 | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/32 | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 12/34 | 14/32 | 13/32 | 9/33
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASN008 1.25% (N=34) | ASN008 2.5% (N=32) | ASN008 5% (N=32) | ASN008 Matching Vehicle (N=33)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Application Site Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema Impetiginous (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Pyuria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heat Exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Creatine Phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood Iron Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Protein Urine Present (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urine Ketone Body Present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine Leukocyte Esterase Positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White Blood Cell Count Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Micturition Urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This trial included an exploratory evaluation of ASN008 pharmacokinetics (PK) as a secondary endpoint using population-based methods. During the analysis, quantifiable levels of ASN008 were unexpectedly observed in vehicle and pre-dose plasma samples. Follow-up investigation indicated this may have been related to assay limitations, which would confound the population PK analysis. Therefore, the analysis was not pursued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT05870865/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT05870865/SAP_001.pdf